CLINICAL TRIAL: NCT01209780
Title: A Multi-center, Phase III, Randomized, Observer Blind Study to Evaluate the Safety, Tolerability and Immunogenicity of a Trivalent Subunit Inactivated Flu Vaccine in Healthy Children and Adolescents 3 to 17 Years of Age
Brief Title: Safety and Immunogenicity of Trivalent Subunit Inactivated Flu Vaccine Administered to Healthy Children and Adolescents 3 to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V71_18
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Seasonal Influenza
Keywords: seasonal influenza, vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- TIV (3-8 years) (Experimental): Non-Naive subjects received one dose and naive subjects received two doses, administered 4 weeks apart, of investigational trivalent influenza vaccine (TIV)
  Interventions: Biological: TIV
- Control TIV (3-8 years) (Active Comparator): Non-Naive subjects received one dose and Naive subjects received two doses, administered 4 weeks apart, of control vaccine. Subjects aged 3 to <4 years and subjects aged 4 to 8 years received different control TIV.
  Interventions: Biological: TIVf; Biological: Comparator TIV
- TIV ( 9-17 years) (Experimental): All subjects received one dose of investigational TIV. The subjects in this cohort were included only for safety analysis.
  Interventions: Biological: TIV
- Control TIV ( (9-17 years) (Active Comparator): All subjects received one dose of the control vaccine. The subjects from this cohort were included only for safety analysis.
  Interventions: Biological: TIVf

INTERVENTIONS:
Biological: TIV — Investigational egg-derived trivalent subunit influenza vaccine.
  Arms: TIV ( 9-17 years); TIV (3-8 years)
Biological: TIVf — US licensed trivalent inactivated subunit influenza vaccine -Fluvirin (Novartis Vaccines and Diagnostics) is approved for use in subjects ≥4 years.
  Arms: Control TIV ( (9-17 years); Control TIV (3-8 years)
Biological: Comparator TIV — US licensed trivalent subunit inactivated influenza vaccine- Fluzone (Sanofi Pasteur) is approved for use in children <4 years.
  Arms: Control TIV (3-8 years)

SUMMARY:
This study will evaluate the safety and immunogenicity in healthy children and adolescents after one or two IM dose(s) of trivalent subunit inactivated flu vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 3 to 17 years, in good health as determined by medical history, physical examination and clinical judgment of the investigator
* Documented consent provided by parents or legal guardians
* For individuals 8 years of age and older, informed assent to participate in the study after the nature of the study had been explained to them in terms they could understand
* Individuals and parents/guardians who were able to comply with all study procedures and were available for all clinic visits scheduled in the study

Exclusion Criteria:

* Parents or legal guardians and individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study
* Parents or legal guardians and individuals providing assent who do not consent to the retention of the subject's serum samples after study completion
* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may have interfered with the subject's ability to participate in the study
* Individuals with history or any illness that, in the opinion of the investigator, might have interfered with the results of the study or posed additional risk to the subjects due to participation in the study
* History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to influenza viral proteins, latex, to any excipients, and to eggs (including ovalbumin), chicken protein, influenza viral protein, kanamycin, neomycin sulphate, cetyltrimethylammonium bromide (CTAB), polysorbate 80, neomycin, polymixin, formaldehyde, thimerosal, beta propiolactone, or nonoxynol-9
* History of any serious disease, such as:

  1. cancer
  2. history of serious chronic, rheumatologic, neurologic and hematologic diseases
  3. history of underlying medical condition such as inborn errors of metabolism
* Known or suspected impairment/alteration of immune function, including:

  1. chronic use of oral steroids within 60 days prior to Visit 1 (use of inhaled, intranasal, or topical corticosteroids is allowed)
  2. receipt of immunostimulants within 60 days prior to Visit 1
  3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within 3 months prior to Visit 1 or planned during the full length of the study
  4. HIV infection or HIV-related disease
* Pregnant or breast-feeding female and any positive or indeterminate pregnancy test
* Received an influenza vaccine within 6 months prior to Visit 1
* Laboratory-confirmed or suspected influenza disease within 6 months prior to Visit 1
* Receipt of another vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study
* Experienced a fever and/or any acute illness within 3 days prior to each study vaccination

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3116 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Centro de Atención e Investigación Medica - CAIMED, Carrera 42A # 17-50, Bogotá, Colombia
- Clinical research institute ,S.C(CRI), Blvd Manuel Avila Camacho 1994 Consultorio 1103 Col. San Lucas Tepetlacalco, C.P.54055 Tlalnepantla, Estado de México, Mexico
- Panama (4):
  - Centro de Salud Magally Ruiz, Street Bolivar, Panama - La Chorrera
  - Clinica Hospital San Fernando, Floor 4 Office 419 via España las Sabanas, Panama City
  - Consultorios America Floor 2 Office 201-1, Via España Vista Hermosa, Panama City
  - Consultorios Medicos San Judas Tadeo Principal Street, Floor 5 Office 507, Villa Lucre, Panama City
- Philippines (7):
  - Philippine General Hospital, Taft Avenue, Manila, Manila
  - Research Institute for Tropical Medicine, Department of Health Compound, Filinvest Corporate City, Alabang, Muntinlupa City
  - Research Institute for Tropical Medicine, Department of Health Compound, FILINVEST Corporate City, Alabang, Muntinlupa City
  - University of the East Ramon Magsaysay Medical Center, 64 Aurora Boulevard, Barangay Dona Imelda Quezon City
  - De La Salle Health Sciences Institute, Dasmarinas Cavite
  - Mary Chiles General Hospital, 667 Gastambide St. Sampaloc, Manila
  - Philippine Children's Medical Center, Quezon Avenue corner Agham Road, Quezon City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 13 centers across 4 countries: Mexico, Colombia, Panama and Philippines.
Pre-assignment Details: Due to GCP non-compliance at the Mexico site, data of 312 subjects (3-8 year olds) enrolled from this site were excluded from the final immunogenicity and safety analysis. The population was analyzed in the enrolled set.
Groups:
- TIV (3-8 Years Old): The group consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination). The non-naive subjects received one dose and naive subjects received two doses of investigational TIV.
- Control (4-8 Years): The group consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination). The non-naive subjects received one dose and naive subjects received two doses of US licensed control vaccine- TIVf.
- Control (3 to < 4 Years): The group consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination.The non-naive subjects received one dose and naive subjects received two doses of US licensed control vaccine- comparator TIV.
- TIV (9-17 Years): All subjects in this group were non-naive and received one dose of investigational TIV.
- Control (9-17 Years): All subjects in this group were non-naive and received one dose of US licensed control vaccine TIVf.
Period: Overall Study
Arm/Group | TIV (3-8 Years Old) | Control (4-8 Years) | Control (3 to < 4 Years) | TIV (9-17 Years) | Control (9-17 Years)
Started | 1042 | 485 | 48 | 817 | 412
Completed | 1016 | 467 | 44 | 807 | 407
Not Completed | 26 | 18 | 4 | 10 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 17 | 12 | 3 | 9 | 4
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Inappropriate enrollment | 0 | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demography reported for all enrolled set except for 312 subjects (3-8 year olds) who were enrolled in the Mexico site.
Groups:
- TIV (3-8 Years): The group consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination). The non-naive subjects received one dose and naive subjects received two doses of investigational TIV.
- Control (3-8 Years): The group [control (4-8 years) + control (3 to<4 years)] consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination). Subjects (4-<9 years) received TIVf and subjects (3-<4 years) received comparator TIV. The non-naive subjects received one dose and naive subjects received two doses of vaccine.
- TIV (9-17 Years): All subjects received one dose of investigational TIV.
- Control (9-17 Years): All subjects received one dose of control TIV (eTIV_f).
- Total: Total of all reporting groups
Arm/Group | TIV (3-8 Years) | Control (3-8 Years) | TIV (9-17 Years) | Control (9-17 Years) | Total
Number analyzed (Participants) | 1042 | 533 | 817 | 412 | 2804
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (1.6) | 5.6 (1.6) | 12.4 (2.4) | 12.3 (2.3) | 8.6 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517 | 269 | 398 | 215 | 1399
  Male | 525 | 264 | 419 | 197 | 1405

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Antibody Responses of Investigational TIV to Control Vaccine in Terms of the Percentage of Subjects Achieving Seroconversion
Description: The non-inferiority of the antibody responses of investigational TIV compared to control TIV assessed in terms of the percentage of subjects achieving seroconversion, against the three homologous vaccine strains,in children 3 to 8 years of age, at 21 days after last vaccination.
  Seroconversion was defined as a pre-vaccination haemagglutinin inhibition (HI) titer <1:10 and post-vaccination HI titer ≥1:40 or as a pre-vaccination HI titer ≥1:10 and at minimum four-fold rise in post-vaccination antibody titer
Time Frame: Day 22 for non-naive/Day 50 for naive subjects
Population: Analysis was done on per protocol population i.e-all subjects who correctly received study vaccinations,provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to unblinding.
Measure: Number (95% Confidence Interval); unit: Percentages
Groups:
- Control (3-8 Years): The group [control (4-8 years) + control (3 to<4 years)] consisted of naive (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) and non-naive subjects (who had a record of previous influenza vaccination). Subjects (4-<9 years) received TIVf and subjects (3-<4 years) received comparator TIV. The non-naive subjects received one dose and naive subjects received two doses of control vaccine.
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 918 | 468
Percentages
  H1N1 strain (N=916,467) | 95 [93 to 96] | 94 [91 to 96]
  H3N2 strain (N=917,468) | 78 [75 to 80] | 87 [84 to 90]
  B strain | 87 [84 to 89] | 85 [82 to 89]
Statistical Analysis 1: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to control TIV against A/H1N1 influenza strain; Test type: Non-Inferiority or Equivalence — The investigational TIV was to be considered non-inferior to the control TIV if for all three strains the upper bound of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion control - Seroconversion investigational) at 21 days after last vaccination does not exceed 10 percentage points; Vaccine group difference (%) = -1, 95% CI 2-sided [-4 to 2]
Statistical Analysis 2: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to control TIV against A/H3N2 influenza strain; Test type: Non-Inferiority or Equivalence — The investigational TIV was to be considered non-inferior to the control TIV if, for all three strains, the upper bound of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion control - Seroconversion investigational), at 21 days after last vaccination, does not exceed 10 percentage points; Vaccine group difference (%) = 10, 95% CI 2-sided [6 to 14]
Statistical Analysis 3: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to the control TIV against B influenza strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Vaccine group difference (%) = -1, 95% CI 2-sided [-5 to 3]

2. Secondary Outcome: Percentages of Subjects Achieving HI Titers ≥40 Following Vaccination With Investigational TIV or Control Vaccine.
Description: The percentages of 3 to 8 year old subjects achieving HI titers ≥40 after receiving either one or two doses of investigational TIV or control vaccine, 21 days after last vaccination, are reported.
  This criterion according to the US (CBER)guideline is met if the lower bound of the two sided 95%CI for percentage of subjects achieving HI titers ≥40, is ≥70%.
Time Frame: Day 22 for non-naive/Day 50 for naive subjects
Population: Analysis was performed on per protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 918 | 468
Percentages of subjects
  Baseline (H1N1strain, N=917,467) | 49 [46 to 53] | 48 [44 to 53]
  Day 22 or Day 50 (H1N1strain; N=917,468) | 97 [95 to 98] | 95 [93 to 97]
  Baseline (H3N2 strain) | 84 [81 to 86] | 85 [82 to 88]
  Day 22 or Day 50 (H3N2 strain; N=917,468) | 100 [100 to 100] | 100 [99 to 100]
  Baseline (B strain) | 23 [21 to 26] | 26 [22 to 30]
  Day 22 or Day 50 (B strain) | 95 [93 to 96] | 92 [90 to 95]

3. Primary Outcome: Comparison of Antibody Responses of Investigational TIV to Control Vaccine in Terms of Post Vaccination Geometric Mean Titers (GMTs)
Description: The non-inferiority of the antibody responses of investigational TIV compared to control vaccine assessed in terms of post vaccination GMTs, at 21 days after last vaccination against the three homologous vaccine strains in 3 to 8 year old children.
Time Frame: Day 22 for non-naive/Day 50 for naive subjects
Population: Analysis was performed on the per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 918 | 468
Titers
  Baseline (H1N1 strain, N=917,467) | 26 [22 to 31] | 28 [25 to 31]
  Day 22 or Day 50 (H1N1 strain,N=917,468) | 1157 [1052 to 1272] | 1501 [1283 to 1756]
  Baseline (H3N2 strain) | 142 [127 to 158] | 150 [129 to 175]
  Day 22 or Day 50 (H3N2 strain, N=917,468) | 1385 [1300 to 1475] | 2032 [1843 to 2240]
  Baseline (B strain) | 12 [11 to 13] | 13 [12 to 14]
  Day 22 or Day 50 (B strain) | 208 [193 to 224] | 195 [174 to 217]
Statistical Analysis 1: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to licensed control TIV against A/H1N1 influenza strain; Test type: Non-Inferiority or Equivalence — The investigational TIV was to be considered non-inferior to the control TIV, if for all three strains, the upper bound of the two-sided 95% CI on the ratio of the GMTs (GMTcontrol/GMTinvestigational) at 21 days after last vaccination does not exceed 1.5; Ratio of GMTs = 1.32, 95% CI 2-sided [1.11 to 1.56]
Statistical Analysis 2: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to licensed control TIV against A/H3N2 influenza strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of GMTs = 1.48, 95% CI 2-sided [1.34 to 1.64]
Statistical Analysis 3: Comparison: TIV (3-8 Years) vs Control (3-8 Years); Non-inferiority of investigational TIV to licensed control TIV against B influenza strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of GMTs = 0.95, 95% CI 2-sided [0.85 to 1.07]

4. Secondary Outcome: Percentages of Subjects With Seroconversion in Antibody Titers Following Vaccination With Investigational TIV or Control Vaccine
Description: The percentages of 3 to 8 years-old subjects achieving seroconversion in HI antibody titers after receiving either one or two doses of investigational TIV or control vaccine, at 21 days after last vaccination, are reported.
  This criterion, according to the US (CBER) guideline, is met if the lower limit of 95% CI of percentage of subjects achieving seroconversion or significant increase at day 22 and day 50 (21 days after last vaccination) is ≥40.
Time Frame: Day 22 for non-naive/Day 50 for naive
Population: Analysis was performed on the per protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 918 | 468
Percentages of subjects
  H1N1 strain (N= 916,467) | 95 [93 to 96] | 94 [91 to 96]
  H3N2 strain ( N= 917,468) | 78 [75 to 80] | 87 [84 to 90]
  B strain | 87 [84 to 89] | 85 [82 to 89]

5. Secondary Outcome: Percentages of Vaccine-naive Children Achieving HI Titers ≥40 After Receiving Two Doses of Investigational TIV or Control Vaccine.
Description: The percentage of 3 to 8 years-old vaccine-naive subjects achieving HI titers ≥40, after receiving two doses of investigational TIV or control vaccine. The time frame of evaluation was 28 days after first (Day 29) and 21 days after second vaccine dose (Day 50).
  This criterion according to the US (CBER) guideline is met if the lower bound of the two sided 95%CI for percentage of subjects achieving HI titers ≥40 is ≥70%, for each vaccine strain.
Time Frame: Day 1, Day 29, and Day 50
Population: Analysis was done on the per protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- TIV (3-8 Years): The group consisted of naive subjects (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) who received two doses of investigational TIV.
- Control (3-8 Years): The group [control (4-8 years) + control (3 to <4 years)] consisted of naive subjects (who have never received influenza vaccination or had received only one influenza vaccine dose in the same season) who received two doses of control vaccine. Subjects (4-<9 years) received TIVf and subjects (3-<4 years) received two doses of comparator TIV.
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 820 | 413
Percentages of subjects
  Day 1 (H1N1 strain, N=819,412) | 49 [46 to 53] | 48 [43 to 53]
  Day 29 (H1N1 strain, N=819,413) | 83 [80 to 86] | 82 [78 to 86]
  Day 50 (H1N1 strain, N= 819,413) | 99 [98 to 100] | 98 [96 to 99]
  Day 1 (H3N2 strain) | 88 [85 to 90] | 90 [87 to 93]
  Day 29 (H3N2 strain, N= 819, 413) | 99 [98 to 100] | 98 [96 to 99]
  Day 50 (H3N2 strain,N= 819, 413) | 100 [100 to 100] | 100 [99 to 100]
  Day 1 (B strain) | 25 [22 to 28] | 26 [22 to 31]
  Day 29 (B strain, N= 820,412) | 82 [79 to 84] | 81 [77 to 85]
  Day 50 (B strain) | 98 [96 to 99] | 94 [92 to 96]

6. Secondary Outcome: Percentages of Vaccine-naive Children Achieving Seroconversion in Antibody Titers, After Receiving Two Doses of Investigational TIV or Control Vaccine
Description: The percentages of 3 to 8 years-old vaccine naive children achieving seroconversion or significant increase in HI antibody titers after receiving two doses of investigational TIV or control vaccine, are reported. The time frame of evaluation was 28 days after first (Day 29) and 21 days after the second dose (Day 50).
  This criterion, according to the US (CBER) guideline, is met if the lower limit of 95% CI of percentage of subjects achieving seroconversion or significant increase at day 29 and day 50 is ≥40, for each vaccine strain.
Time Frame: Day 29 and Day 50
Population: Analysis was done on the per protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV (3-8 Years) | Control (3-8 Years)
Number analyzed (Participants) | 820 | 413
Percentages of subjects
  Day 29 (H1N1 strain, N= 818,412) | 82 [79 to 84] | 81 [77 to 85]
  Day 50 (H1N1 strain, N= 818,412) | 98 [96 to 99] | 96 [94 to 98]
  Day 29 (H3N2 strain, N= 819,413) | 74 [71 to 77] | 87 [83 to 90]
  Day 50 (H3N2 strain, N= 819,413) | 78 [75 to 80] | 87 [84 to 90]
  Day 29 (B strain, N= 820,412) | 74 [71 to 77] | 73 [68 to 77]
  Day 50 (B strain) | 89 [87 to 91] | 88 [85 to 91]

7. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events After Vaccination With Investigational TIV and Control Vaccine
Description: The number of 3-17 year old children with solicited local and systemic adverse events and other adverse events, after receiving either one or two doses of investigational TIV as compared to control vaccine are reported.
Time Frame: Day 1 to 7 after vaccination
Population: Analysis was done on the safety set population i.e all subjects who received at least one study vaccine and provided post vaccination safety data.
Measure: Number; unit: Subjects
Groups:
- Control (9-17 Years): All subjects received one dose of control vaccine(TIVf).
Arm/Group | TIV (3-8 Years) | Control (3-8 Years) | TIV (9-17 Years) | Control (9-17 Years)
Number analyzed (Participants) | 1037 | 531 | 817 | 412
Subjects
  Any local | 364 | 216 | 270 | 148
  Injection site pain | 363 | 215 | 268 | 146
  Injection site ecchymosis | 1 | 1 | 2 | 0
  Injection site erythema | 1 | 1 | 2 | 1
  Injection site induration | 10 | 6 | 5 | 6
  Injection site swelling | 11 | 11 | 6 | 3
  Any systemic | 262 | 161 | 193 | 94
  Chills | 37 | 20 | 38 | 8
  Malaise | 77 | 51 | 68 | 27
  Myalgia | 78 | 50 | 54 | 34
  Arthralgia | 41 | 20 | 26 | 12
  Headache (N=1037,531,817,411) | 101 | 52 | 93 | 38
  Sweating | 37 | 29 | 43 | 22
  Fatigue | 34 | 22 | 52 | 21
  Fever (≥ 38°C) | 116 | 68 | 39 | 12
  Other | 153 | 89 | 103 | 54
  Analgesic/Antipyretic med.used(N=1032,531,816,412) | 91 | 52 | 22 | 9
  Stayed at home due to reaction(N=1019,524,809,411) | 93 | 54 | 89 | 49

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Vaccination With Investigational TIV and Control Vaccine
Description: The number of 3-17 year old children reporting any unsolicited adverse event and any serious adverse event (SAE) after receiving either one or two doses of investigational TIV and control vaccine are reported.
Time Frame: Day 1 to 180 (non-naive )/Day 1 to 209 (naive)
Population: Analysis was done on the safety set population.
Measure: Number; unit: Subjects
Groups:
- Control (9-17 Years): All subjects received one dose of control vaccine (TIVf).
Arm/Group | TIV (3-8 Years) | Control (3-8 Years) | TIV (9-17 Years) | Control (9-17 Years)
Number analyzed (Participants) | 1039 | 531 | 817 | 412
Subjects
  Any adverse event | 395 | 194 | 101 | 58
  At least possibly related adverse event | 64 | 36 | 23 | 11
  Serious adverse event | 14 | 3 | 4 | 3
  At least possibly related serious adverse event | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events collected from Day 1-7 after each vaccination. Serious adverse events and other unsolicited adverse events were collected from Day 1-180 for non-naive and Day 1-209 for vaccine-naive subjects.
Description: The population analyzed here is the safety set.
Groups:
- Control (9-17 Years): All subjects received one dose of control vaccine (TIV_f).
Arm/Group | TIV (3-8 Years) | Control (3-8 Years) | TIV (9-17 Years) | Control (9-17 Years)
Serious Adverse Events (participants affected / at risk) | 14/1039 | 3/531 | 4/817 | 3/412
Other Adverse Events (participants affected / at risk) | 657/1039 | 342/531 | 385/817 | 196/412
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIV (3-8 Years) (N=1039) | Control (3-8 Years) (N=531) | TIV (9-17 Years) (N=817) | Control (9-17 Years) (N=412)
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Ascariasis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cholera (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Measles (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIV (3-8 Years) (N=1039) | Control (3-8 Years) (N=531) | TIV (9-17 Years) (N=817) | Control (9-17 Years) (N=412)
injection site pain (General disorders) | 363 | 215 | 268 | 146
malaise (General disorders) | 77 | 52 | 68 | 27
pyrexia (General disorders) | 164 | 91 | 43 | 15
nasopharingitis (Infections and infestations) | 85 | 37 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 102 | 41 | 0 | 0
fatigue (General disorders) | 0 | 0 | 52 | 21
myalgia (Musculoskeletal and connective tissue disorders) | 79 | 51 | 54 | 34
headache (Nervous system disorders) | 106 | 54 | 94 | 41
hyperhidrosis (Skin and subcutaneous tissue disorders) | 37 | 29 | 43 | 22

LIMITATIONS AND CAVEATS:
Due to GCP non-compliance at the Mexico site, data of 312 subjects (3-8 year olds) enrolled from this site were excluded from the final immunogenicity and safety analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days